CLINICAL TRIAL: NCT03559166
Title: A Phase Ia/Ib, Randomized, Double Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of BLD-2660 in Healthy Volunteers and Patients With Lung Fibrosis or Liver Fibrosis
Brief Title: First in Human Study in Healthy Volunteers Followed With Dosing in Participants With Lung or Liver Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blade Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-2660-101
Record Dates: First submitted 2018-04-24; First posted 2018-06-18 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Fibrosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, double-blind, placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- cohort 1a - starting dose (Experimental): Single oral dose of BLD-2660 or placebo capsule administered to healthy volunteers
  Interventions: Drug: BLD-2660
- cohort 1b- first SAD escalation (Placebo Comparator): Single oral dose of BLD-2660 or placebo capsule(s) administered to healthy volunteers (1st dose escalation)
  Interventions: Drug: BLD-2660
- cohort 1c-2nd SAD escalation (Placebo Comparator): Single oral dose of BLD-2660 or placebo capsule(s) administered to healthy volunteers (2nd dose escalation) in fasting state, followed by washout period and then single oral dose of BLD-2660 or placebo administered to healthy volunteers in fed state.
  Interventions: Drug: BLD-2660
- cohort 1d-3rd SAD escalation (Placebo Comparator): Single oral dose of BLD-2660 or placebo capsules(s) administered to healthy volunteers (3rd dose escalation)
  Interventions: Drug: BLD-2660
- cohort 1e-4th SAD escalation (Placebo Comparator): Single oral dose of BLD-2660 or placebo capsule(s) administered to healthy volunteers (final dose escalation if assessed as safe).
  Interventions: Drug: BLD-2660
- cohort 2a-1st MAD cohort (Placebo Comparator): Multiple oral doses of BLD-2660 or placebo capsule(s) administered to healthy volunteers
  Interventions: Drug: BLD-2660
- cohort 2b-2nd MAD escalation (Placebo Comparator): Multiple oral doses of BLD-2660 or placebo capsule(s) administered to healthy volunteers.
  Interventions: Drug: BLD-2660
- cohort 2c-3rd MAD escalation (Placebo Comparator): Multiple oral doses of BLD-2660 or placebo capsule(s) administered to healthy volunteers.
  Interventions: Drug: BLD-2660
- cohort 2d-4th MAD escalation (Placebo Comparator): Multiple oral doses of BLD-2660 or placebo capsule(s) administered to healthy volunteers.
  Interventions: Drug: BLD-2660
- cohort 2e-5th MAD escalation (Placebo Comparator): Multiple oral doses of BLD-2660 or placebo capsule(s) administered to healthy volunteers.
  Interventions: Drug: BLD-2660
- cohort 2F-6th MAD escalation (Placebo Comparator): Multiple oral doses of BLD-2660 or placebo capsule(s) administered to healthy volunteers.
  Interventions: Drug: BLD-2660

INTERVENTIONS:
Drug: BLD-2660 — Randomized to active product or placebo
  Other Names: Placebo

SUMMARY:
First in Human single ascending dose followed by multiple ascending doses in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Agree to no smoking or alcohol or illegal substance 48 hours prior to dosing
* Have a negative urine drug screen/alcohol breath test on admission to clinic
* Agree to use highly effective, double barrier contraception (both male and female partners) during the study and for 30 days following completion of dosing
* Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1
* Normal BMI except liver fibrosis participants (BMI 18 to ≤35 kg/m2)
* Be in general good health
* Clinical laboratory values within normal range
* Lung fibrosis participants-a diagnosis of lung fibrosis,
* Liver fibrosis participants-a diagnosis of liver fibrosis; some abnormal laboratory values will be acceptable for the following; platelet count, albumin, serum creatinine and neutrophil-leukocyte ration

Exclusion Criteria:

* Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the subject will complete the study per protocol
* History or presence of alcoholism or drug abuse within the 2 years prior to the first study drug administration, and unwillingness to be totally abstinent during the dosing period
* Blood donation or significant blood loss within 60 days prior to the first study drug administration
* Plasma donation within 7 days prior to the first study drug administration
* Administration of investigational product (IP) in another trial within 30 days prior to the first study drug administration, or five half-lives, whichever is longer
* Females who are pregnant or lactating
* Surgery within the past 3 months prior to the first study drug administration determined by the PI to be clinically relevant
* Failure to satisfy the PI of fitness to participate for any other reason
* Active infection or history of recurrent infections
* Active malignancy and history of malignancy in the past 5 years, with the exception of completely excised basal cell carcinoma or low grade cervical intraepithelial neoplasia
* Chronic obstructive pulmonary disease
* Antibiotic treatment within 3 months
* Chronic medical condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 2 weeks
  AEs will be assessed by determining the incidence, severity, and dose relationship of adverse events
Any observed changes in clinical safety laboratory results | 2 weeks
  Assessed by reviewing any observed changes in CBC, serum chemistry or urinalysis from baseline by dose. Results in subjects dosed with BLD-2660 treatment will be compared to those dosed with placebo.
Any observed changes in physical examinations | 2 weeks
  Assessed by reviewing any observed changes in physical examinations from baseline by dose. Results in subjects dosed with BLD-2660 will be compared to those dosed with placebo.
Any observed changes in vital signs | 2 weeks
  Assessed by reviewing any observed changes in vital signs from baseline by dose. Results in subjects dosed with BLD-2660 will be compared to those dosed with placebo.
Any observed changes in ECG | 2 weeks
  Assessed by reviewing any observed changes in ECG from baseline by dose. Results in subjects dosed with BLD-2660 will be compared to those dosed with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Snyder, MD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia